CLINICAL TRIAL: NCT06473298
Title: EFFICACY OF VISUAL LIGHT TRACKING ON CHILDREN WITH SPASTIC HEMIPLEGIA
Brief Title: Role of Light Tracking Intervention in Children With Spastic Hemiplegia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, MAHMOUD AHMED GOUDA ALI ABDELAZIZ ABDELMONEIM, Bachelor's degree in Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Light Tracking in Hemiplegia
Record Dates: First submitted 2024-06-07; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Spastic Hemiplegic Cerebral Palsy
Keywords: Visual Light Tracking

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual light tracking program (Experimental): Visual light tracking program
  Interventions: Other: Visual Light Tracking
- Selective physical therapy program (Experimental): Selective physical therapy program
  Interventions: Other: Visual Light Tracking

INTERVENTIONS:
Other: Visual Light Tracking — visual light tracking program consists of 10 tasks every task lasts for 6 minutes and may be repeated for the child especially in the first sessions to give him trials to him/her to understand the exercise.

SUMMARY:
The study aims to investigate the effect of visual light tracking on gait, selective motor control and sensory processing in children with spastic hemiplegic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from (4-7 years).
* They will be able to walk independently.
* They will have intact auditory pathways.
* They will have intact visual pathways.
* They will have a mild degree of spasticity graded from 1 to 1+ according to the modified Ashworth scale
* They will be mentally stable.

Exclusion Criteria:

* Any other neuromuscular disorders.
* Convulsion.
* Botox injection
* Fixed deformities of lower limbs and spine.
* Selective dorsal rhizotomy (SDR).
* Children with spasticity more than 1+ according to the modified Ashworth scale.
* Children with visual disorders such as squint myopia.
* children with auditory problems.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Effect of Visual light tracking intervention on quality of walking, selective motor control and sensory processing of the study group compared to control group with different intervention. | Baseline
  The quality of walking as step length will be assessed using Kinovea software. Selective motor control will be assessed using Selective Control Assessment of the Lower Extremity (points).
  Sensory processing will be assessed using the Sensory Proﬁle Caregiver Questionnaire(points).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt